CLINICAL TRIAL: NCT04670406
Title: A Guided Online Acceptance and Commitment Therapy (ACT) Intervention Combined With Psychoeducation for People With Spinal Cord Injury: A Preliminary Study
Brief Title: A Guided Online ACT Intervention Combined With Psychoeducation for People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Areum Han, Assistant professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006536
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Spinal Cord Injuries; Psychological Distress
Keywords: Acceptance and Commitment Therapy; Quality of life; Spinal cord injury; Psychological distress; Depression; Anxiety; Stress; Mindfulness; Self-compassion
MeSH Terms: conditions — Spinal Cord Injuries; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acceptance and commitment therapy (ACT) combined with psychoeducation (Experimental): Participants receive 8 weekly sessions, including 6 ACT sessions and 2 psychoeducation sessions, delivered by trained coaches through Zoom videoconferencing.
  Interventions: Behavioral: acceptance and commitment therapy (ACT) combined with psychoeducation

INTERVENTIONS:
Behavioral: acceptance and commitment therapy (ACT) combined with psychoeducation — Participants receive 8 weekly sessions, including 6 ACT sessions and 2 psychoeducation sessions, delivered by trained coaches through Zoom videoconferencing.

SUMMARY:
The purpose of this preliminary study is to examine the effects of a guided online acceptance and commitment therapy (ACT) intervention combined with psychoeducation on people with spinal cord injury (SCI) who experience psychological distress.

DETAILED DESCRIPTION:
This project will employ a one-group pretest-posttest design to investigate the effects of a guided online acceptance and commitment therapy (ACT) intervention combined with psychoeducation on quality of life and mental health of people with spinal cord injury (SCI) who experience psychological distress. After the pretest evaluation, eligible participants will receive 8 weekly sessions, including 6 ACT sessions and 2 psychoeducation sessions, delivered by trained coaches through Zoom videoconferencing. Each session lasts for one hour. Primary outcome measures will be psychological distress measured by the Depression, Anxiety and Stress Scale (DASS)- 21 and Spinal Cord Injury - Quality of Life (SCI-QOL). A one-time interview at the completion of the 8 sessions will be conducted to explore participants' experiences in the sessions.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults (age 18 or over) living in the community who had a spinal cord injury
* suffering at least mild symptoms of psychological distress measured by the DASS-21
* having a computer/smartphone with internet access capable of doing web browsing and video-conferencing
* being able to provide informed consent by understanding the nature of study participation.

Exclusion Criteria:

* having cognitive, physical, or sensory deficits, or language barriers (non- English communicator) that impede study participation
* receiving a psychological therapy currently
* having psychiatric hospitalizations or diagnoses of mental illness in the previous 2 years
* taking antipsychotic or anticonvulsant medication at the time of recruitment
* having the possibility of study dropouts due to other medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS) - 21 | Change from baseline to 8 weeks
  The Depression, Anxiety and Stress Scale (DASS)- 21 is a 21-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and stress. Higher scores represent greater symptomatology.
World Health Organization Quality of Life Instruments (WHOQOL-BREF) - psychological health component | Change from baseline to 8 weeks
  WHOQOL-BREF - psychological health component has 6 items measuring: bodily image and appearance; negative feelings; positive feelings; self-esteem; spirituality / personal beliefs; and thinking, learning, memory and concentration. Higher scores denote higher quality of life in terms of psychological health.

SECONDARY OUTCOMES:
Self-Compassion Scale- Short Form (SCS-SF) | Change from baseline to 8 weeks
  Self-Compassion Scale- Short Form (SCS-SF) has 12 items assessing the relation of self-compassion to positive psychological health. Higher scores indicate higher levels of self-compassion.
Engagement in Meaningful Activities Survey (EMAS) | Change from baseline to 8 weeks
  The Engagement in Meaningful Activities Survey (EMAS) is a 12-item self-assessment instrument that measures a person's subjective experience of the meaningfulness of everyday activities. Higher scores indicate greater levels of engagement in meaningful activities.
Action and Acceptance Questionnaire (AAQ)-II | Change from baseline to 8 weeks
  The Action and Acceptance Questionnaire (AAQ)-II is a 7-item self-report questionnaire measuring psychological flexibility. Higher scores indicate poor psychological flexibility.
Cognitive Fusion Questionnaire (CFQ)-7 | Change from baseline to 8 weeks
  The Cognitive Fusion Questionnaire (CFQ)-7 is a 7-item self-report questionnaire measuring cognitive fusion. Higher scores indicate greater levels of cognitive fusion.
Spinal Cord Injury - Quality of Life (SCI-QOL) Grief and Loss Short form | Change from baseline to 8 weeks
  SCI-QOL Grief and Loss Short form has 9 items assessing grief and loss due to spinal cord injuries. Higher scores indicate more grief/loss.
Spinal Cord Injury - Quality of Life (SCI-QOL) Resilience Short form | Change from baseline to 8 weeks
  SCI-QOL Resilience Short form has 8 items assessing resilience. Higher scores indicate more resilience.
Mindful Attention Awareness Scale (MAAS) | Change from baseline to 8 weeks
  The MAAS is a 15-item scale assessing dispositional mindfulness (i.e., open or receptive awareness of and attention to what is taking place in the present). Higher scores reflect higher levels of dispositional mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han A, Wilroy JD, Jenkins J, Yuen HK. Effects of a coach-guided videoconferencing acceptance and commitment therapy intervention combined with psychoeducation on distressed individuals living with spinal cord injury: a preliminary mixed-methods study. Disabil Rehabil. 2023 Feb;45(4):644-654. doi: 10.1080/09638288.2022.2038283. Epub 2022 Feb 12. PMID 35156500